CLINICAL TRIAL: NCT01830348
Title: A Randomized, Double-blind, Parallel-group, Vehicle-controlled Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of DSC127 in Treating Non-healing Foot Ulcers in Subjects With Diabetes Mellitus
Brief Title: Phase III Study to Evaluate Efficacy and Safety of DSC127 in Diabetic Foot Ulcers
Acronym: STRIDE 1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSC127-2012-01
Record Dates: First submitted 2013-03-15; First posted 2013-04-12 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Diabetic Foot Ulcers
Keywords: diabetic foot ulcers; Wagner Grade 1 or 2 foot ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — aclerastide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DSC127 (Active Comparator): DSC127 0.03% in a vehicle gel (hydroxyethyl cellulose (HEC) with parabens)
  Interventions: Drug: DSC127
- Vehicle gel (Placebo Comparator): Vehicle gel comprising HEC with parabens
  Interventions: Drug: placebo vehicle gel

INTERVENTIONS:
Drug: DSC127 — DSC127 0.03%, daily topical application to diabetic foot ulcer for a period of up to 28 days or until ulcer closure, whichever is sooner
  Arms: DSC127
Drug: placebo vehicle gel
  Arms: Vehicle gel

SUMMARY:
The purpose of the study is to determine if DSC127 is effective in increasing incidence of complete wound closure at 10 weeks confirmed at a visit 2 weeks later when compared to the vehicle (gel without active ingredient) in subjects with diabetes mellitus (DM) who have chronic Wagner Grade 1 or 2 plantar neuropathic foot ulcers, 0.75 - 6 cm2 in size.

DETAILED DESCRIPTION:
Subjects will undergo a two week screening period to assess plantar ulcer healing, and those healing less than 30% will be eligible for randomization, providing they meet all other inclusion criteria. Four weeks of blinded "treatment" follows the screening period, and an observation period of six weeks (to 10 weeks post first treatment) follows the 4-week treatment period. If the ulcer closes during the treatment or observation period, the closure will be confirmed two weeks later, and at this time the subject enters a durability assessment period of up to 12 weeks.

All aspects of Standard of Care are followed throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ambulatory subject age ≥18 years at the time of informed consent
2. Has type 1 or type 2 DM under metabolic control as confirmed by a glycosylated hemoglobin (HbA1c) of ≤12% and a serum creatinine level of ≤3mg/dL
3. At Screening and at Baseline (prior to randomization), subject has at least one ulcer that fulfills all of the following criteria:

   * Present for ≥1 month and ≤1 year
   * Partial- or full- thickness and not involving bone, tendon, or capsule (probing to tendon or capsule), i.e. Wagner Grade 1 or 2
   * Has no sign of infection or osteomyelitis
   * Plantar neuropathic ulcer; ulcer must be predominantly on the plantar surface of the foot to ensure adequate off-loading and may include the toes
   * Size of the target ulcer must be 0.75 - 6 cm2
   * Target ulcer must be non-healing as defined as <30% reduction in size in response to standard of care during the two week Screening Period

     * If more than one ulcer is present that meets the inclusion criteria, the largest one will be considered the Target ulcer.
     * If there are two ulcers of the same size that meet all criteria, the one with the higher Wagner Grade will be considered the Target ulcer.
     * If there are two ulcers of the same size and the same Wagner Grade, the one present for the longest qualifying time will be the Target ulcer.
4. Has an ankle brachial index (ABI) ≥ 0.7 on the foot with the target ulcer
5. Has an assessment of the baseline level of neuropathy of the foot using Semmes-Weinstein filaments.
6. A female subject of childbearing potential must have a negative serum pregnancy test at the time of Screening, and must be willing to use a medically acceptable method of birth control, such as Essure®, hormonal contraception (oral pills, implantable device, or skin patch), intrauterine device, tubal ligation, or double barrier throughout the study. A female subject of childbearing potential who practices abstinence is not required to employ birth control.
7. Has the ability and willingness to understand and comply with study procedures and to give written informed consent prior to enrollment in the study or initiation of study procedures

Exclusion Criteria:

1. Has a known hypersensitivity to any of the investigational drug or vehicle components
2. Has been exposed to any investigational agent within 30 days of entry into the study
3. A female who is pregnant or nursing
4. Has active malignant disease of any kind except for basal cell carcinoma (of the skin). A subject, who has had a malignant disease in the past, was treated and is currently disease-free, may be considered for study entry.
5. Has a hemoglobin of less than 8.5 gm/dL.
6. Transaminase levels greater than 3 × normal
7. Is receiving hemodialysis or chronic ambulatory peritoneal dialysis (CAPD) therapy
8. Has had prior radiation therapy of any part of the foot with the target ulcer under study
9. Use of systemic corticosteroids and immunosuppressants (within the 8 weeks prior to screening)
10. Has an ulcer primarily ischemic in etiology
11. Has sickle-cell anemia, Reynaud's, or other peripheral vascular disease
12. Has received a biologic agent, growth factors or skin equivalents (Regranex®, Apligraft, or Dermagraft), in the past 30 days
13. Has a target ulcer which is determined to be clinically infected and requires antimicrobials. Any antibiotic therapy must be completed or discontinued at screening.
14. Has a Wagner Grade 3 or greater DFU, deep abscess, or gangrene
15. Has uncontrolled hypertension, in the opinion of the Investigator.
16. Any other finding, which in the opinion of the Investigator, may interfere with the assessment of the product or participation of the subject in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with a target ulcer which achieves complete wound closure (skin re-epithelialization without drainage or dressing requirements) up to 10 weeks (confirmed at a study visit 2 weeks later). | Target ulcer must achieve complete wound closure by 10 weeks post first treatment
  Primary endpoint of complete closure is assessed by the Principal Investigator at the site; ulcer measurements are calculated through tracings submitted to the Canfield system and photographs are collected as confirmation of closure via the Canfield system.

SECONDARY OUTCOMES:
Time to the visit where the target ulcer achieves confirmed complete wound closure | Weekly assessments to ten weeks post first treatment dose

OTHER OUTCOMES:
Percent reduction in ulcer area per week (closure rate) | Weekly ulcer tracings to calculate area of ulcer, measurements continue to ten weeks post first treatment dose
  Calculated weekly for up to ten weeks
Incidence of target ulcer recurrence, time to ulcer recurrence, and number of days target ulcer remains closed after confirmed complete wound closure has been established. | Assessed during a 12 week durability period following the confirmation of complete wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Gere S diZerega, MD, Study Director — Integra LifeSciences Corporation
Locations (25):
- United States (25):
  - WILMAX Clinical Research Inc, Mobile, Alabama
  - Center for Clinical Research, Fair Oaks, California
  - Roy O Kroeker, DPM, Inc, Fresno, California
  - Foot and Ankle Clinic, Los Angeles, California
  - Brian O'Carroll, DPM, Inc., Pismo Beach, California
  - UCLA Medical Center - Olive View, Sylmar, California
  - Orange County Research Center, Tustin, California
  - Advanced Research Institute of Miami, Homestead, Florida
  - UF Health Orthopaedic Surgery Clinic, Jacksonville, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - GF Professional Research, Miami Lakes, Florida
  - Barry University Clinical Research, North Miami Beach, Florida
  - Professional Health Care of Pinellas, St. Petersburg, Florida
  - Memorial Medical Group, Granger, Indiana
  - LaPorte Medical Group, La Porte, Indiana
  - Boston University Medical Center, Boston, Massachusetts
  - East Carolina Foot and Ankle Specialists, Greenville, North Carolina
  - Clinical Research Center, Eugene, Oregon
  - Center for Clinical Research, Portland, Oregon
  - Carolina Musculoskeletel Institute, Aiken, South Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - Fort Worth Diagnostic Clinic, Fort Worth, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Professional Education and Research Institute, Roanoke, Virginia